CLINICAL TRIAL: NCT03634384
Title: Rapid Use of High-sensitive Cardiac Troponin I for ruling-in and Ruling-out of Acute Myocardial Infarction
Acronym: RACING-MI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Bo Løfgren, Professor, MD, PhD, FESC, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: 54559
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Myocardial Infarction; Chest Pain
Keywords: Myocardial Infarction; Chest Pain
MeSH Terms: conditions — Myocardial Infarction; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Lithium-Heparin, Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation cohort: We include eligible patients presenting with chest pain suggestive of myocardial infarction to the emergency department (see eligibility).
  For the primary study patients will be divided into two groups: 500 patients will serve as derivation cohort.
- Validation cohort: We include eligible patients presenting with chest pain suggestive of myocardial infarction to the emergency department (see eligibility).
  For the primary study patients will be divided into two groups: 500 patients will serve as validation cohort.

SUMMARY:
Early rule-in or rule-out of myocardial infarction (MI) is essential in patients presenting to the Emergency Department with chest pain. Recently, the European Society of Cardiology has suggested an accelerated 0h/1h algorithm to rule-in or rule-out MI as a valid alternative to the standard 0h/3h approach. So far, the 0h/1h algorithm has only been validated for certain high-sensitive Troponin assays. Moreover, it is unknown if MI can be ruled-out by measuring hs-cTn already at 30 minutes (0h/30m) after presentation to the Emergency Department.

This prospective cohort study aims to investigate, if a high-sensitive Troponin assay can rule-in or rule-out MI, when using a 0h/30m and a 0h/1h algorithm. Serial blood samples will be drawn from each patient and used for biomarker analysis. In addition, patients will be asked to complete a detailed questionnaire on chest pain characteristics.

DETAILED DESCRIPTION:
Background: Chest pain is a key symptom of acute coronary syndrome (ACS), but can also represent other cardiac and non-cardiac diseases. Rapid identification of ACS in terms of 'rule-in' or 'rule-out' is essential in order to minimize treatment delay and time to discharge. In the absence of ST-segment elevation myocardial infarction (STEMI) at initial ACS evaluation, the European Society of Cardiology guidelines recommend repeated measurements of high-sensitive cardiac troponin (hs-cTn) at presentation (0h) and 3 hours (3h) after presentation to rule-in and rule-out myocardial infarction (MI). An accelerated algorithm for ruling-in and ruling-out MI after 1h (0h/1h algorithm) has recently been suggested by the European Society of Cardiology as a valid alternative to the standard approach. The novel 0h/1h algorithm has only been validated for certain hs-cTn assays. However, routine use of the 0h/1h algorithm is still not widely implemented, as further data on algorithm performance are warranted.

A study of patients undergoing transcoronary ablation of septal hypertrophy, a clinical model of MI, shows that troponin concentrations measured by a hs-cTn assay significantly increase already after 15 minutes. This indicates that it may be possible to evaluate troponin dynamics even earlier than suggested by the 0h/1h algorithm. So far, no large-scale studies have included measurements of hs-cTn at 30m, and no 0h/30m algorithm has been derived. Therefore it is unknown if rule-in and rule-out of MI can be done safely using a 0h/30m algorithm.

Aim: To investigate if a high-sensitive Troponin Assay can rule-in or rule-out MI, when using a 0h/30m and a 0h/1h algorithm.

Patients and methods: This prospective cohort study will include patients presenting to the Emergency Department with chest pain suggestive of ACS. The study is designed to enroll 1.000 patients with complete blood samples (0h, 30m, 1h and 3h).

The expected incidence of MI in our population is inevitably low due to pre-hospital risk-stratification based on point-of-care troponin and electrocardiogram evaluation in the ambulance. Thus, patients with a very high pre-test probability of MI will be admitted to tertiary care centers with cardiac catheterization facilities rather than a regional hospital as in present study. Pilot study calculations estimate an expected prevalence of MI in our study cohort of approximately 7.4%. Assuming a negative predictive value of 99.7% in the rule-out group, a distribution with 7% patients in the rule-in group and 20% assigned to the observational zone (patients who can't be stratified to either the rule-out or the rule-in group), enrolment of at least 500 patients for derivation of the algorithms and at least 500 for the validation of the respective algorithms will provide an acceptable lower boundary of 98.2% of the two-sided 95% confidence interval.

All patients aged ≥18 years referred to the emergency department at Randers Regional Hospital, Randers, Denmark with chest pain and admitted on the suspicion of ACS will be eligible for the study. Patients will be recruited after initial contact with an emergency department nurse when results of an electrocardiogram as well as vital sign parameters (blood pressure, heart rate, peripheral oxygen saturation, respiratory rate and temperature) are available. Patients <18 years of age, with STEMI at admission, in dialysis treatment or pregnant will be excluded.

The study is conducted in accordance with the Declaration of Helsinki. Oral and written consent will be obtained. Patients will be asked for informed consent to have information passed on from the electronic patient journal regarding gender, age, medicine, previous MI and co-morbidity for use in this study only. Patients declining to participate will receive standard treatment.

Serial blood samples will be drawn at 0h (admission), 30m, 1h and 3h. The blood samples will be analyzed using high-sensitive troponin assays. Additional blood will be stored for each time point to establish a research biobank. Troponin values and troponin dynamics will be paired with final diagnosis for each patient. Two independent physicians will adjudicate the patients' final diagnosis based on data from the electronic patient journal (including physical examination, patient history, laboratory results, electrocardiogram, and other examinations). In cases of disagreement, a consensus decision will be reached after a case review. The treating physician will be blinded to test results at 30m and 1h, with the final therapeutic decision being left to the discretion of the attending physician and relying on troponin measurements at 0h and 3h only. All patients will be asked to complete a questionnaire on, e.g., time of chest pain onset and peak, chest pain characteristics (localization, radiation, sensation), additional symptoms at presentation (diaphoresis, nausea, abdominal pain, syncope, dyspnoea, palpitations), height and weight, smoking status and family history of coronary artery disease.

Significance: This study challenges existing time limits for ACS evaluation by investigating the diagnostic value of hs-cTnI measurements at 30m. If our study shows that rule-out of MI can be performed safely at 30m, ACS evaluation can potentially be accelerated even further. Furthermore, our study will provide data on the performance of the 0h/1h algorithm in a Danish patient cohort. If this study demonstrates that the 0h/1h diagnostic algorithm can be used to safely rule-out MI in a patient cohort with a different risk profile, it can contribute to the acceptance of novel accelerated diagnostic approaches and favor global implementation of the 0h/1h algorithm.

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years of age
* Admitted to the Emergency Department
* Chest pain suggestive of myocardial infarction.

Exclusion criteria:

* Patients <18 years of age
* STEMI at admission
* Dialysis
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain suggestive of myocardial infarction admitted to the Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of the 0h/1h algorithm in terms of ruling-out MI. | 1 hour after admission blood samples
  The negative predictive value of the 0h/1h algorithm
The diagnostic performance of the 0h/30m algorithm in terms of ruling-out MI. | 30 minutes after admission blood samples
  The negative predictive value of the 0h/30m algorithm

SECONDARY OUTCOMES:
Overall diagnostic performance of the 0h/1h algorithm. | 1 hour after admission blood samples
  The positive predictive value, sensitivity and specificity of the 0h/1h algorithm.
Overall diagnostic performance of the 0h/30m algorithm. | 30 minutes after admission blood samples
  The positive predictive value, sensitivity and specificity of the 0h/30m algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Løfgren, Professor, MD, PhD, Study Director — Randers Regional Hospital; Camilla Bang, MD, Principal Investigator — Randers Regional Hospital; Camilla Hansen, MD, Principal Investigator — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohn JK, Cohn PF. Cardiology patient pages. Chest pain. Circulation. 2002 Jul 30;106(5):530-1. doi: 10.1161/01.cir.0000027208.17824.d6. No abstract available. PMID 12147530
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Jaeger C, Wildi K, Twerenbold R, Reichlin T, Rubini Gimenez M, Neuhaus JD, Grimm K, Boeddinghaus J, Hillinger P, Nestelberger T, Singeisen H, Gugala M, Pretre G, Puelacher C, Wagener M, Honegger U, Schumacher C, Moreno Weidmann Z, Kreutzinger P, Krivoshei L, Freese M, Stelzig C, Dietsche S, Ernst S, Rentsch K, Osswald S, Mueller C. One-hour rule-in and rule-out of acute myocardial infarction using high-sensitivity cardiac troponin I. Am Heart J. 2016 Jan;171(1):92-102.e1-5. doi: 10.1016/j.ahj.2015.07.022. Epub 2015 Jul 26. PMID 26699605
- [Background] Reichlin T, Schindler C, Drexler B, Twerenbold R, Reiter M, Zellweger C, Moehring B, Ziller R, Hoeller R, Rubini Gimenez M, Haaf P, Potocki M, Wildi K, Balmelli C, Freese M, Stelzig C, Freidank H, Osswald S, Mueller C. One-hour rule-out and rule-in of acute myocardial infarction using high-sensitivity cardiac troponin T. Arch Intern Med. 2012 Sep 10;172(16):1211-8. doi: 10.1001/archinternmed.2012.3698. PMID 22892889
- [Background] Reichlin T, Twerenbold R, Wildi K, Gimenez MR, Bergsma N, Haaf P, Druey S, Puelacher C, Moehring B, Freese M, Stelzig C, Krivoshei L, Hillinger P, Jager C, Herrmann T, Kreutzinger P, Radosavac M, Weidmann ZM, Pershyna K, Honegger U, Wagener M, Vuillomenet T, Campodarve I, Bingisser R, Miro O, Rentsch K, Bassetti S, Osswald S, Mueller C. Prospective validation of a 1-hour algorithm to rule-out and rule-in acute myocardial infarction using a high-sensitivity cardiac troponin T assay. CMAJ. 2015 May 19;187(8):E243-E252. doi: 10.1503/cmaj.141349. Epub 2015 Apr 13. PMID 25869867
- [Background] Mueller C, Giannitsis E, Christ M, Ordonez-Llanos J, deFilippi C, McCord J, Body R, Panteghini M, Jernberg T, Plebani M, Verschuren F, French J, Christenson R, Weiser S, Bendig G, Dilba P, Lindahl B; TRAPID-AMI Investigators. Multicenter Evaluation of a 0-Hour/1-Hour Algorithm in the Diagnosis of Myocardial Infarction With High-Sensitivity Cardiac Troponin T. Ann Emerg Med. 2016 Jul;68(1):76-87.e4. doi: 10.1016/j.annemergmed.2015.11.013. Epub 2016 Jan 12. PMID 26794254
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members; Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):2354-94. doi: 10.1161/CIR.0000000000000133. Epub 2014 Sep 23. No abstract available. PMID 25249586
- [Background] Liebetrau C, Mollmann H, Nef H, Szardien S, Rixe J, Troidl C, Willmer M, Hoffmann J, Weber M, Rolf A, Hamm C. Release kinetics of cardiac biomarkers in patients undergoing transcoronary ablation of septal hypertrophy. Clin Chem. 2012 Jun;58(6):1049-54. doi: 10.1373/clinchem.2011.178129. Epub 2012 Apr 13. PMID 22504118
- [Derived] Andersen CF, Bang C, Lauridsen KG, Frederiksen CA, Schmidt M, Jensen T, Hornung N, Lofgren B. External validation of a high-sensitive troponin I algorithm for rapid evaluation of acute myocardial infarction in a Danish cohort. Eur Heart J Acute Cardiovasc Care. 2021 Dec 6;10(9):1056-1064. doi: 10.1093/ehjacc/zuab062. PMID 34423355
- [Derived] Andersen CF, Bang C, Lauridsen KG, Frederiksen CA, Schmidt M, Jensen T, Hornung N, Lofgren B. Single troponin measurement to rule-out acute myocardial infarction in early presenters. Int J Cardiol. 2021 Oct 15;341:15-21. doi: 10.1016/j.ijcard.2021.08.005. Epub 2021 Aug 13. PMID 34391791
- [Derived] Bang C, Hansen C, Lauridsen KG, Frederiksen CA, Schmidt M, Jensen T, Hornung N, Lofgren B. Rapid use of high-sensitive cardiac troponin I for ruling-in and ruling-out of acute myocardial infarction (RACING-MI): study protocol. Open Heart. 2019 Apr 3;6(1):e000995. doi: 10.1136/openhrt-2018-000995. eCollection 2019. PMID 31168384

DOCUMENTS (1):
  • Study Protocol (2018-08-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT03634384/Prot_000.pdf